CLINICAL TRIAL: NCT03593499
Title: Expanded Access to Omaveloxolone for Melanoma for Patients Previously Enrolled in 408-C-1401
Status: No longer available | Type: Expanded Access
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 408-C-1401EA
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Melanoma
Keywords: melanoma; omaveloxolone; expanded access
MeSH Terms: conditions — Melanoma | interventions — omaveloxolone

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: omaveloxolone
  Other Names: RTA 408

SUMMARY:
This is an expanded access program for eligible participants and is designed to provide access to omaveloxolone for the treatment of unresectable or metastatic melanoma to patients who previously participated in the 408-C-1401 (REVEAL) study. To be considered for expanded access, a Principal Investigator from the REVEAL trial should submit a request to Reata Pharmaceuticals on behalf of the individual patient.

DETAILED DESCRIPTION:
Study Sponsor, originally Reata Pharmaceuticals, Inc., is now Reata Pharmaceuticals, Inc., a wholly owned subsidiary of Biogen.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult